CLINICAL TRIAL: NCT03695692
Title: Assistant Professor, Physioterapist, PhD
Brief Title: Effects of Connective Tissue Massage in Women With Overactive Bladder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seyda TOPRAK CELENAY (Other)
Responsible Party: Sponsor-Investigator, Seyda TOPRAK CELENAY, Assistant Professor, Ataturk Training and Research Hospital
Organization: Ataturk Training and Research Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/07-01
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connective tissue massage group (Experimental): Pelvic floor exercises and connective tissue massage have been applied
  Interventions: Behavioral: pelvic floor exercise and connective tissue massage
- Control group (Experimental): Pelvic floor exercises alone have been applied
  Interventions: Behavioral: pelvic floor exercise

INTERVENTIONS:
Behavioral: pelvic floor exercise and connective tissue massage — Pelvic floor exercises with connective tissue massage will be performed.The massage program is carried out for 18 sessions, 3 days/week in 6 weeks. The exercise program is performed every day for 6 weeks
  Arms: Connective tissue massage group
Behavioral: pelvic floor exercise — The exercise program is performed every day for 6 weeks
  Arms: Control group

SUMMARY:
The aim of this study was to compare the effects of pelvic floor muscle trainig with connective tissue massage and only pelvic floor muscle training in women with overactive bladder

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age,
* having overactive bladder
* being volunteer

Exclusion Criteria:

* being in the period of pregnancy or breastfeeding,
* having an accompanying neurological disease, presence of a mental issue that would prevent cooperation in examinations and/or implementations, history of acute infectionor presence of a malignce

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
overactive bladder symptoms measured by Overactive Bladder Questionnaire_V8 | Change from baseline bladder symptoms at 6 weeks
  Overactive Bladder Questionnaire_V8 assessing severity of overactive bladder symptoms will be used. This scale includes items on urgency, incontinence, nocturia and voiding frequency, as defined by the International Continence Society, referring to the previous four weeks. The final score is the sum of the partial scores obtained for each of the eight questions, ranging from 0 to 40. Patients with a final score of eight or more are considered as having Overactive Bladder symptoms.

SECONDARY OUTCOMES:
urgency complaint assessed with The patient's Perception of Intensity of Urgency Scale | Change from baseline urgency complaints at 6 weeks
  The patient's Perception of Intensity of Urgency Scale assessing urgency complaints will be used. This scale is scored on 0 and 4 points (the best score is '0' and the worst score is '4') based on urgency complaints. Higher scores indicate more severe urgency complaints.
quality of life assessed with King's Health Questionnaire (KHQ) | Change from baseline quality of life at 6 weeks
  King's Health Questionnaire assessing quality of life related to urinary problems will be used. This questionnaire consists of two parts and 32 items. The first part (21 items) contains two single-item questions that address General Health Perception and Incontinence Impact and the following seven multi-item domains: Role, Physical, and Social Limitations, Limitations in Personal Relationship, Emotional Problems, Sleep and Energy Disturbances associated with UI, and Severity Measures for UI. The second part has an 11-item Symptom Severity Scale (SSS) that assesses the presence and severity of urinary symptoms. While the entire SSS is scored from 0 (best) to 30 (worst), the minimum possible score is 0 (best health) and the maximum possible score is 100 (worst health) for all other KHQ domains.
pelvic floor muscle strength measured with perineometer | Change from baseline pelvic floor muscle strength at 6 weeks
  change in pelvic floor muscle strength as measued with perineometer
diurnal urinary frequency, nocturia, maximum urinary volume, the number of urinary leakage and pad changes measured with voiding dairy | Change from baseline diurnal urinary frequency, nocturia, maximum urinary volume, the number of urinary leakage and pad changes at 6 weeks
  Patients will be also instructed to keep voiding diary for three days. In this diary, diurnal urinary frequency, nocturia, maximum urinary volume, the number of urinary leakage and pad changes will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Seyda TOPRAK CELENAY, Principal Investigator — Ankara Yildirim Beyazıt University; Yasemin Karaaslan, Study Chair — Beykent University; Faruk Kucukdurmaz, Study Chair — Kahramanmaras Sutcu Imam University
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Turkey (Türkiye)